CLINICAL TRIAL: NCT01575821
Title: The Effect of Honey on Nocturnal Cough and Sleep Quality: a Double-blind, Randomized,Placebo-controlled Study
Brief Title: The Effect of Honey on Nocturnal Cough and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Collaborators: Ambulatory Pediatric Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: hermanhoney
Record Dates: First submitted 2012-04-08; First posted 2012-04-12 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Cough; Sleep
Keywords: children, cough, honey
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Eucalyptus honey , (Experimental): 75 children
  Interventions: Dietary Supplement: Eucalyptus honey
- Labiatae honey (Experimental): 75 children allocated
  Interventions: Dietary Supplement: Labiatae honey
- Silan date extract (placebo) (Experimental): 75 children allocated
  Interventions: Dietary Supplement: Silan date extract
- Citrus honey (Experimental): 75 children allocated
  Interventions: Dietary Supplement: Citrus honey

INTERVENTIONS:
Dietary Supplement: Eucalyptus honey — Parents were instructed to administer 10 grams of theirs child treatment product (single dose) within 30 minutes of the child going to sleep.
  Arms: Eucalyptus honey ,
Dietary Supplement: Labiatae honey — Parents were instructed to administer 10 grams of theirs child treatment product (single dose) within 30 minutes of the child going to sleep.
  Arms: Labiatae honey
Dietary Supplement: Citrus honey — Parents were instructed to administer 10 grams of theirs child treatment product (single dose) within 30 minutes of the child going to sleep.
  Arms: Citrus honey
Dietary Supplement: Silan date extract — Parents were instructed to administer 10 grams of theirs child treatment product (single dose) within 30 minutes of the child going to sleep.
  Arms: Silan date extract (placebo)

SUMMARY:
Cough is a common symptom in pediatric practice. It can be particularly troubling to children and their parents.It often results in discomfort to the child and loss of sleep to both the child and the parent. The objective of this trial was to compare the effects on nocturnal cough and the sleep difficulty associated with URIs of a single nocturnal dose of three different honey products compared to placebo

DETAILED DESCRIPTION:
Cough is a common symptom in pediatric practice.As a result, children miss daycare or school and parents miss a day of work. In an attempt to threat cough, caregivers frequently administer OTC medication to their children,with their attendant risks, kack of proven efficacy and the disapproval of professional organizations such as the AAP and the FDA. The WHO has noted honey as a potential treatment for cough and cold symptoms. Honey has antioxidant properties and increases cytokine release. The objective of this trial was to compare the effects on nocturnal cough and the sleep difficulty associated with URIs of a single nocturnal dose of three different honey products compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* 1-5 years of age complying of nocturnal cough that was attributed to a URI.

Exclusion Criteria:

* asthma,
* pneumonia,
* laryngotracheobronchitis,
* sinusitis,
* allergic rhinitis,
* use of cough or cold medication on the night before entering the study.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2009-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The principal outcome measure of interest was the change in the frequency of cough between the 2 nights (before treatment and tthe night with treatment). | changes between two nights ( the night before treatment and the night with treatment)
  Pre intervention study questionnaire:
  The parents were asked to complete a five item questionnaire regarding parental subjective assessments of the child's cough and sleep difficulty on the previous night.Survey responses were graded on a seven point scale ranging from extremely (6 points) to not at all (0 points). On the day following the treatment,the parent completed the same questionnaire that had been answered before the intervention, this time regarding the previous evening when the child had received the treatment.

SECONDARY OUTCOMES:
changes in the cough severity, the bothersome nature of the cough, the effect of the cough on sleep for both the child and parents between the two nights | changes between two nights ( the night before treatment and the night with treatment)
  Assessment was been done by completing the pre and post intervention questionnaire as was described in the " primary outcome measurment".

CONTACTS AND LOCATIONS:
Overall Officials: Cohen AV Herman, Principal Investigator — Israel Clalit Health Services
Locations (1):
- 6 General Pediatric Community Clinics, Petah Tikva, Israel

REFERENCES:
- [Background] Paul IM, Beiler J, McMonagle A, Shaffer ML, Duda L, Berlin CM Jr. Effect of honey, dextromethorphan, and no treatment on nocturnal cough and sleep quality for coughing children and their parents. Arch Pediatr Adolesc Med. 2007 Dec;161(12):1140-6. doi: 10.1001/archpedi.161.12.1140. PMID 18056558
- [Derived] Cohen HA, Rozen J, Kristal H, Laks Y, Berkovitch M, Uziel Y, Kozer E, Pomeranz A, Efrat H. Effect of honey on nocturnal cough and sleep quality: a double-blind, randomized, placebo-controlled study. Pediatrics. 2012 Sep;130(3):465-71. doi: 10.1542/peds.2011-3075. Epub 2012 Aug 6. PMID 22869830